CLINICAL TRIAL: NCT03936855
Title: Clinical Evaluation of Posterior Direct Restoration in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Renata Afonso da Silva Pereira (Other)
Collaborators: Coordination for the Improvement of Higher Education Personnel (Other); Fundação de Amparo à Pesquisa do estado de Minas Gerais (Other); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Sponsor-Investigator, Renata Afonso da Silva Pereira, PHD student, Federal University of Uberlandia
Organization: Federal University of Uberlandia (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UFU001
Record Dates: First submitted 2019-05-01; First posted 2019-05-03 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Composite Resins

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Incremental filling technique (Active Comparator): Glass ionomer in the pulp chamber and incremental filling technique using composite resin
  Interventions: Procedure: Direct composite resin
- Bulk Fill (Experimental): Bulk fill composite resin filling all the cavity
  Interventions: Procedure: Direct composite resin

INTERVENTIONS:
Procedure: Direct composite resin — For both groups: The teeth will have the enamel surface conditioned with 37% phosphoric acid. For the restorative procedure, the same adhesive system will be used
  GROUP ACTIVE COMPARATOR
  1. Insert resin-modified glass ionomer cement into the pulp chamber;
  2. Complete the restoration by incremental technique using conventional composite resin in increments of 2mm;
  EXPERIMENTAL GROUP
  1. Insert Bulk Fill composite inside the pulp chamber to the height of 5 mm;
  2. Complete the insertion of the Bulk Fill resin to the limit of the caval surface angle in the occlusal

SUMMARY:
The present study aims to evaluate the performance of direct restorations with bulk fill resins in molars with great structural loss, with endodontic treatment. The behavior of class II restorations in 68 molars endodontically treated with bulk fill resin and incremental technique will be evaluated by means of a randomized clinical trial with a two-year follow-up. This project aims to evaluate the performance of this new restorative strategy that can greatly contribute to restorations of posterior teeth.

DETAILED DESCRIPTION:
Sixty-eight endodontically treated molars were restored in 54 adolescents (10-18 years old, mean= 14.0 +- 2.4). Teeth were randomly assigned to the incremental filling technique (Filtek Z230/Vitremer, 3M-ESPE, n = 31) or high viscosity bulk fill technique (Filtek Bulk Fill Posterior, 3M-ESPE, n = 37). The restorations were clinically evaluated at baseline, 12 and 24 months by two independent raters using modified United States Public Health Service criteria. Data analysis included descriptive statistics, Mann-Whitney and Friedman non-parametric tests, and Generalized Estimating Equation (GEE) analysis.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents with necessity of endodontic treatment in molar teeth, to be aged between 10 and 18 years;
* Patients that require direct restorations in Class II MOD cavities in molar teeth;
* Patients with medical history that does not compromise the evolution of the results;
* Patients that have a habit of oral hygiene involving brushing teeth at least once a day;
* Patients that have normal periodontal condition against the probing parameters.

Exclusion Criteria:

* Patients with some chronic disease with oral manifestations;
* Patients who present some serious oral pathology;
* Patients with no oral hygiene;
* Patients with allergies to any material that will be used on this study;
* Patients presenting with signs or symptoms of bruxism and dental tightening;
* Patients with teeth that will be used as a pillar for removable prosthesis or fixed partial dentures;
* Patients with teeth with porcelain restorations directly opposite the tooth that will receive the restoration.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 54 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
restoration failure | 2 years
  material fraction

SECONDARY OUTCOMES:
marginal staining | 2 years
  color alteration in the adhesive interface

CONTACTS AND LOCATIONS:
Overall Officials: Carlos J Soares, DDS,MS,PHD, Study Chair — Universidade Federal de Uberlândia
Locations (1):
- Universidade Federal de Uberlândia, Uberlândia, Minas Gerias, Brazil

IPD SHARING:
Plan to Share IPD: No